CLINICAL TRIAL: NCT00808938
Title: A Pilot Study of the Use of Magnetic Seizure Therapy for Treatment Resistant Depression
Brief Title: A Pilot Study of the Use of Magnetic Seizure Therapy for Depression
Acronym: MST
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bayside Health (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 28508
Record Dates: First submitted 2008-12-15; First posted 2008-12-16 (Estimated); Last update posted 2013-02-13 (Estimated); Status verified 2008-12

CONDITIONS: Treatment Resistant Depression
MeSH Terms: conditions — Depressive Disorder, Treatment-Resistant

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Active Treatment (Experimental)
  Interventions: Device: MST

INTERVENTIONS:
Device: MST — Magnetic Seizure Therapy

SUMMARY:
Electro convulsive therapy (ECT) remains the only established therapy for the large percentage of patients with depression who fail to respond to standard treatments. It is commonly used but has substantial problems including the occurrence of cognitive side effects that are often highly distressing for patients. The development of a new treatment with similar efficacy but which minimises these side effects would have great clinical value. One highly promising possibility is magnetic seizure therapy (MST). MST involves replacing the electrical stimulation used in ECT with a magnetic stimulus. This appears to be able to produce similar clinical effects but without the disabling cognitive side effects related to ECT. However, substantive trials using the newest MST equipment are required. Due to the rarity of the equipment available so far, these are only being undertaken in a handful of places internationally and no research with MST has occurred in Australia. The investigators are fortunate to have been able to obtain one of the very limited number of MST devices available internationally and are proposing a pilot study of this technique. Conduct of a successful pilot study would be strong justification for an application for a large head-to-head MST - ECT comparison trial. Should MST be shown to have similar efficacy to ECT but with reduced side-effects, it is envisioned that it could rapidly replace ECT in clinical practice throughout Australia and indeed internationally with substantial ongoing benefits to patients. These would include enhanced use of it as an outpatient therapy as well as the reduction in side-effects.

The study will be an open label trial of MST in 15 patients with treatment resistant depression who have been referred for ECT. All patients will undergo a dose titration procedure to establish seizure threshold, six MST treatment sessions will then be provided at 120% of threshold. If the patients have not achieved a 50% reduction in their depressive symptoms (as measured by the Montgomery Asberg Depression Rating Scale rating scale) patients will receive another 12 sessions. MST will be administered three times a week. Patients will undergo a series of assessments to determine both the efficacy of MST and the cognitive outcomes. The primary outcome measure will be the MADRS measure of depression severity. The investigators will additionally measure patient rated depression severity and cognitive functioning The overall aim of the current project is to, via an open label pilot trial, investigate the clinical response to magnetic seizure therapy in patients with treatment resistant depression who have been referred for electroconvulsive therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Have a DSM-IV diagnosis of a major depressive episode
2. Are referred for or an outpatient course of ECT at the Alfred Hospital
3. Age 18-75
4. Have a Montgomery-Asberg Depression Rating Scale (MADRS) score of > 25 (moderate - severe depression)
5. Demonstration of capacity to give informed consent: this will be assessed by the study psychiatrist as well as the patient's primary treating psychiatrist.

Exclusion Criteria:

1. Have an unstable medical condition, or neurological disorder or are currently pregnant or lactating.
2. Patients not considered sufficiently well to undergo general anaesthesia for any reason
3. Patients with cardiac pacemakers, cochlear implants or other implanted electronic devices. Patients with non-electric metallic implants will also be excluded.
4. Significant concurrent axis 1 or 11 psychiatric comorbidity.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2009-01; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
MADRS | 2 weeks

SECONDARY OUTCOMES:
Cognitive Assessment | 2 - 6 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Alfred Psychiatry Research Centre, Prahran, Victoria, Australia

REFERENCES:
- [Derived] Fitzgerald PB, Hoy KE, Herring SE, Clinton AM, Downey G, Daskalakis ZJ. Pilot study of the clinical and cognitive effects of high-frequency magnetic seizure therapy in major depressive disorder. Depress Anxiety. 2013 Feb;30(2):129-36. doi: 10.1002/da.22005. Epub 2012 Oct 18. PMID 23080404